CLINICAL TRIAL: NCT07159100
Title: Neuromodulation as a Therapeutic Intervention to Improve Cancer Related Fatigue and Weakness
Brief Title: tDCS for Cancer-Related Fatigue and Weakness
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Guang Yue, Director, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R 1012-18
Record Dates: First submitted 2025-08-15; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Cancer-related Fatigue; Neuromodulation
Keywords: tDCS; Cancer-related fatigue; neuromodulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS (Experimental): 1.5-2.0 mA stimulation over motor cortex during fatigue task.
  Interventions: Device: Active tDCS + elbow flexion exercise
- Sham tDCS (Sham Comparator): Stimulation for 30 seconds with ramping to mimic active sensation.
  Interventions: Drug: Sham tDCS + elbow flexion exercise

INTERVENTIONS:
Device: Active tDCS + elbow flexion exercise — Participants will receive anodal tDCS targeting motor-related cortical areas using either traditional sponge-based or high-definition (HD)-tDCS configurations. The intervention is delivered at 1.5-2.0 mA for 20-30 minutes, either before or during a sustained submaximal isometric contraction task designed to induce fatigue.
  tDCS will be administered in a counterbalanced crossover design, where each participant completes both active stimulation and sham stimulation conditions in separate sessions spaced at least one week apart. Sham stimulation mimics the sensory effects of active tDCS (30-second ramp-up and down) without delivering sustained current.
  The intervention is unique as the target population is cancer survivors with persistent fatigue >6 months post-treatment. Also, the tDCS is combined with neurophysiological assessments, including EMG, TMS, EEG, and MRI, to provide neurophysiological evidence of acute effects.
  Other Names: Active tDCS
  Arms: Active tDCS
Drug: Sham tDCS + elbow flexion exercise — Participants will receive anodal tDCS targeting motor-related cortical areas using either traditional sponge-based or high-definition (HD)-tDCS configurations. The intervention is delivered at 1.5-2.0 mA for 30 seconds to mimic the sensation of active tDCS (20 minutes long), either before or during a sustained submaximal isometric contraction task designed to induce fatigue.
  tDCS will be administered in a counterbalanced crossover design, where each participant completes both active stimulation and sham stimulation conditions in separate sessions spaced at least one week apart. Sham stimulation mimics the sensory effects of active tDCS (30-second ramp-up and down) without delivering sustained current.
  Arms: Sham tDCS

SUMMARY:
This pilot study investigates the effectiveness of non-invasive brain stimulation (tDCS) in alleviating cancer-related fatigue (CRF) and muscle weakness. Using a randomized, double-blind crossover design, participants perform fatiguing muscle tasks with and without tDCS, and outcomes include task endurance, maximal voluntary contraction force, and neuromuscular markers. Neural mechanisms will be assessed via EEG, TMS, and MRI.

ELIGIBILITY:
General Inclusion - All participants

1. Aged 40-80
2. Right Handed, as determined by the Edinburgh Inventory 21
3. Proficient in English
4. Must be available for the familiarization, and testing sessions

General Inclusion - Cancer Patients only

1. Cancer (>6 months post therapy)
2. Suffers from a subjective feeling of cancer related fatigue and weakness as assessed by the following question: "Do you suffer from symptoms of fatigue and weakness related to your cancer or cancer treatment?"
3. Have had cancer diagnosis and treatment in the past
4. Must have a stable physical/health condition for the past 3 months with no expected changes for the duration of the study

General Exclusion - All participants

1. Neurological, psychiatric, musculoskeletal or other types of disorder not caused by cancer and/or cancer treatment, which may affect participants sensorimotor function and cognitive abilities
2. No consciousness to understand and sign informed consent voluntarily
3. History of alcohol, and illicit drug use
4. History of smoking within the last 5 years.

General Exclusion - Cancer Patients 1. Radiation, surgery, chemo, or other cancer treatment therapies in the past 6 months prior to enrollment. Hormonal maintenance treatment is allowed.

General Exclusion - Healthy Participants

1. History of cancer or cancer treatment

Exclusion criteria related to tDCS and TMS safety - All participants

1. History of epilepsy or unprovoked seizures
2. Family history of epilepsy (father, mother, children, siblings with diagnosis of epilepsy)
3. Active migraine headaches
4. Past or current history of treated tinnitus or severe hearing problems
5. Implanted medical devices (pacemakers, defibrillators, medical pump, implanted brain stimulator, aneurysm clip, carotid or cerebral stents, central venous catheter, non-removable hearing aids)
6. Damage to the skin on the scalp
7. History of mental illness (schizophrenia, anxiety, major depression, manic disorders)
8. Tattoo with metal based ink in the head or neck
9. Currently taking or withdrawing from any central nervous system active medication (stimulants, anticonvulsants, antidepressants, psychotropic medications).
10. Pregnant as determined by a Pregnancy test for non-menopausal (no menstruation for at least 1 year) women younger than 55 years (for TMS and fMRI only).

Exclusion criteria related to MRI safety - All participants

We will be using the Kessler Foundation RONIC MRI center screening form to screen participants for the MRI scan. Exclusion criteria includes:

1. Suffer from claustrophobia (fear of confined spaces)
2. Prior injury to the eye involving a metallic object or fragment (e.g., metallic slivers, shavings, foreign body, etc.)?
3. Presence or prior injury by a metallic object, or foreign body or metallic fragment (e.g., BB, bullet, shrapnel, etc.)
4. Currently or former metal worker (welder, machinist, etc.)
5. Implanted electrical devices (e.g. pacemakers, defibrillators or ICD)
6. Implanted stimulators or internal electrodes or wires (neurostimulator, brain stimulator, spinal cord, bone growth/bone fusion)
7. Aneurysm clips (metal clips on the wall of a large artery), metallic stent, shunt (spinal)
8. Metallic prostheses or implants (including metal pins and rods, plate, screw, surgical staples, clips or metallic sutures, joint replacement (hip, knee), cochlear or other otologic implant, eye, penile, heart valves, eyelid spring or wires, prosthetic limbs)
9. Dental implants, dentures or partial plates (regular filling, amalgam and crown are OK)
10. Insulin, medication or other infusion pumps
11. Radiation seeds or implants
12. Transdermal medication patch (Nitroglycerine, Nicotine)
13. IUD, diaphragm or pessary
14. Tissue expander (e.g. breast)
15. Body tattoos or permanent makeup (eyeliner, lip) if deemed unsafe in the MRI
16. Body piercing

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue task duration | Immediately post-intervention in each experimental session.
  Duration (in seconds) that participants are able to maintain a submaximal isometric contraction (20-40% of maximal voluntary contraction) during a fatigue-inducing task, performed with and without transcranial direct current stimulation (tDCS).
Muscle Strength | Immediately after each stimulation session
  Peak muscle force (in Newtons) generated during a maximal voluntary contraction (MVC) of the arm muscles, assessed immediately before and after the fatiguing isometric contraction task. Comparison is made across active tDCS and sham conditions to determine the acute effects of neuromodulation on post-fatigue strength. Force is measured using a calibrated force sensor.

SECONDARY OUTCOMES:
EMG root mean squared amplitude | Immediately after each stimulation session
  RMS amplitude of surface EMG signals recorded from elbow flexor muscles during the fatigue task. This metric quantifies neuromuscular activity and is used to assess the change in motor unit recruitment from the start to the end of the fatiguing task. EMG is acquired concurrently with force data and compared across tDCS and sham sessions.
Interpolated Twitch Force (Peripheral Fatigue Index) | Immediately after each stimulation session
  Amplitude (in Newtons) of superimposed twitch responses elicited by peripheral nerve stimulation at regular intervals during the fatigue task. This measure assesses muscle reserve and peripheral fatigue by comparing twitch force amplitude pre- and post-task. A reduction in twitch force reflects greater peripheral contribution to fatigue.
Motor Evoked Potential (MEP) Amplitude | Immediately after each stimulation session
  Amplitude (in µV) of motor evoked potentials (MEPs) recorded via surface EMG in response to single-pulse TMS over the motor cortex. MEPs are measured at baseline and post-fatigue to assess changes in corticospinal excitability, and are compared across stimulation conditions (tDCS vs sham) and participant groups (cancer vs healthy controls)
EEG Functional Connectivity | Immediately after each stimulation session
  Change in EEG functional connectivity within the motor network (primary motor cortex, premotor, supplementary motor, and somatosensory cortices) from pre- to post-fatigue states. EEG is recorded using a 64-channel cap and analyzed using EEGLAB-based pipelines to quantify connectivity changes via measures such as coherence or phase-locking value.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Yue, PhD, Study Director — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States